CLINICAL TRIAL: NCT02098395
Title: A 26-weeks Randomised, Insulin Capped, Placebo-controlled, Double-blind, Parallel Group, Multinational, Multi-centre Trial
Brief Title: The Efficacy and Safety of Liraglutide Adjunct to Insulin Treatment in Type 1 Diabetes
Acronym: ADJUNCT TWO™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9211-4083; 2012-005778-74 (EudraCT Number); U1111-1138-0619 (Other: WHO); NL47705.060.14 (Registry Identifier: CCMO); REec-2014-0884 (Registry Identifier: Spanish registry)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Liraglutide 1.8 mg + insulin (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide 1.2 mg + insulin (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide 0.6 mg + insulin (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide placebo 0.3 ml + insulin (Placebo Comparator)
  Interventions: Drug: placebo
- Liraglutide placebo 0.2 ml + insulin (Placebo Comparator)
  Interventions: Drug: placebo
- Liraglutide placebo 0.1 ml + insulin (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Subjects randomised to 1.8 mg liraglutide treatment as an add-on to their pre-trial insulin treatment will receive 0.6 mg liraglutide for 2 weeks followed by 1.2 mg liraglutide for 2 weeks. After 4 weeks of treatment subjects will receive 1.8 mg liraglutide for 22 weeks. Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide 1.8 mg + insulin
Drug: liraglutide — Subjects randomised to 1.8 mg liraglutide treatment as an add-on to their pre-trial insulin treatment will receive 0.6 mg liraglutide for 2 weeks followed by 1.2 mg liraglutide for 2 weeks. After 4 weeks of treatment subjects will receive 1.8 mg liraglutide for 22 weeks. Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide 1.2 mg + insulin
Drug: liraglutide — Subjects randomised to 1.8 mg liraglutide treatment as an add-on to their pre-trial insulin treatment will receive 0.6 mg liraglutide for 2 weeks followed by 1.2 mg liraglutide for 2 weeks. After 4 weeks of treatment subjects will receive 1.8 mg liraglutide for 22 weeks. Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide 0.6 mg + insulin
Drug: placebo — Subjects randomised to 0.3 mL liraglutide placebo as an add-on to their pre-trial insulin treatment will receive 0.1 mL for 2 weeks followed by 0.2 mL for 2 weeks. After 4 weeks of liraglutide placebo, subjects will receive 0.3 mL for 22 weeks. Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide placebo 0.3 ml + insulin
Drug: placebo — Subjects randomised to 0.3 mL liraglutide placebo as an add-on to their pre-trial insulin treatment will receive 0.1 mL for 2 weeks followed by 0.2 mL for 2 weeks. After 4 weeks of liraglutide placebo, subjects will receive 0.3 mL for 22 weeks. Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide placebo 0.2 ml + insulin
Drug: placebo — Subjects randomised to 0.3 mL liraglutide placebo as an add-on to their pre-trial insulin treatment will receive 0.1 mL for 2 weeks followed by 0.2 mL for 2 weeks. After 4 weeks of liraglutide placebo, subjects will receive 0.3 mL for 22 weeks. Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide placebo 0.1 ml + insulin

SUMMARY:
This trial is conducted in Africa, Europe and North America. The purpose of the trial is to investigate the efficacy and safety of liraglutide adjunct to insulin treatment in type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, aged equal to or greater than 18 years at the time of signing informed consent
* Type 1 diabetes mellitus (as diagnosed clinically) 12 months or longer prior to Visit 1 (i.e. screening)
* Treatment with basal bolus or CSII (continuous subcutaneous insulin infusion, insulin pump) treatment 6 months or longer prior to Visit 1 (i.e. screening)
* Stable insulin treatment 3 months or longer prior to Visit 1 (i.e. screening), as judged and documented by the investigator
* HbA1c 7.0-10.0 percent (Diabetes Control and Complications Trial (DCCT)), both inclusive, by central laboratory analysis (Visit 1, screening) corresponding to 53-86 mmol/mol (International Federation of Clinical Chemistry (IFCC))

Exclusion Criteria:

* Prior use of glucagon-like peptide-1 (GLP-1) receptor agonist or dipeptidyl peptidase IV (DPPIV) inhibitors
* Use of any medication, which in the investigator's opinion could interfere with the glycaemic control (e.g. systemic corticosteroids, pramlintide (Symlin®)) or affect the subject's safety. Premix insulin is not allowed
* Known proliferative retinopathy or maculopathy requiring acute treatment
* Severe neuropathy, in particular autonomic neuropathy, i.e. gastroparesis, as judged by the investigator
* Uncontrolled/untreated blood pressure at screening (Visit 1) (after resting for 5 minutes) while sitting greater than 160 mmHg for systolic or greater than 100 mmHg for diastolic (repeated measurement at Visit 2 (prior to performing the trial related activities) is allowed to exclude white-coat hypertension)
* History of acute or chronic pancreatitis
* Screening (Visit 1) calcitonin value equal to or greater than 50 ng/L

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 835 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (116):
- United States (46):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Maitland, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Champaign, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Jamaica, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Murray, Utah
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Bennington, Vermont
  - Novo Nordisk Investigational Site, Federal Way, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Seattle, Washington
- Austria (2):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Vienna
- Belgium (9):
  - Novo Nordisk Investigational Site, Aalst
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Boussu
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Kortrijk
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Mouscron
  - Novo Nordisk Investigational Site, Sint-Niklaas
- Bulgaria (5):
  - Novo Nordisk Investigational Site, Blagoevgrad
  - Novo Nordisk Investigational Site, Pazardzhik
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Razgrad
  - Novo Nordisk Investigational Site, Sofia
- Canada (9):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Cornwall, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Thornhill, Ontario
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
- Denmark (4):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Odense
- Finland (6):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Joensuu
  - Novo Nordisk Investigational Site, Jyväskylä
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Pori
  - Novo Nordisk Investigational Site, Turku
- France (10):
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Pierre-Bénite
  - Novo Nordisk Investigational Site, Reims
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Trinité - La Martinique
- Italy (7):
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Sesto San Giovanni (MI)
  - Novo Nordisk Investigational Site, Siena
- Netherlands (6):
  - Novo Nordisk Investigational Site, 's-Hertogenbosch
  - Novo Nordisk Investigational Site, Amersfoort
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Utrecht
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Spain (4):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Gijón
  - Novo Nordisk Investigational Site, Segovia
  - Novo Nordisk Investigational Site, Seville
- Sweden (6):
  - Novo Nordisk Investigational Site, Ängelholm
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Umeå

REFERENCES:
- [Result] Ahren B, Hirsch IB, Pieber TR, Mathieu C, Gomez-Peralta F, Hansen TK, Philotheou A, Birch S, Christiansen E, Jensen TJ, Buse JB; ADJUNCT TWO Investigators. Efficacy and Safety of Liraglutide Added to Capped Insulin Treatment in Subjects With Type 1 Diabetes: The ADJUNCT TWO Randomized Trial. Diabetes Care. 2016 Oct;39(10):1693-701. doi: 10.2337/dc16-0690. Epub 2016 Aug 4. PMID 27493132
- [Result] Hoogenhout M, Malcolm-Smith S. Theory of mind predicts severity level in autism. Autism. 2017 Feb;21(2):242-252. doi: 10.1177/1362361316636758. Epub 2016 Aug 19. PMID 27493232
- [Derived] Shah VN, Agesen RM, Bardtrum L, Christiansen E, Snaith J, Greenfield JR. Determinants of Liraglutide Treatment Discontinuation in Type 1 Diabetes: A Post Hoc Analysis of ADJUNCT ONE and ADJUNCT TWO Randomized Placebo-Controlled Clinical Studies. J Diabetes Sci Technol. 2025 Mar;19(2):321-331. doi: 10.1177/19322968241305647. Epub 2024 Dec 24. PMID 39717993
- [Derived] Dejgaard TF, von Scholten BJ, Christiansen E, Kreiner FF, Bardtrum L, von Herrath M, Mathieu C, Madsbad S; ADJUNCT ONE and ADJUNCT TWO Investigators. Efficacy and safety of liraglutide in type 1 diabetes by baseline characteristics in the ADJUNCT ONE and ADJUNCT TWO randomized controlled trials. Diabetes Obes Metab. 2021 Dec;23(12):2752-2762. doi: 10.1111/dom.14532. Epub 2021 Sep 28. PMID 34463425
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomised at 113 sites in 13 countries: Austria 2 sites, Belgium 9 sites, Bulgaria 5 sites, Canada 9 sites, Denmark 4 sites, Finland 6 sites, France 9 sites, Italy 7 sites, Netherlands 5 sites, South Africa 2 sites, Spain 5 sites, Sweden 5 sites, United States 45 sites.
Groups:
- Liraglutide 0.6 mg: Subjects randomised to 0.6 mg liraglutide treatment as an add-on to their pre-trial insulin treatment and remained on this dose throughout the trial (26 weeks). Administered subcutaneously (s.c., under the skin) once daily.
- Liraglutide 1.2 mg: Subjects randomised to 1.2 mg liraglutide treatment as an add-on to their pre-trial insulin treatment received 0.6 mg liraglutide for 2 weeks followed by 1.2 mg liraglutide for 24 weeks. Administered subcutaneously (s.c., under the skin) once daily.
- Liraglutide 1.8 mg: Subjects randomised to 1.8 mg liraglutide treatment as an add-on to their pre-trial insulin treatment received 0.6 mg liraglutide for 2 weeks followed by 1.2 mg liraglutide for 2 weeks. After 4 weeks of treatment subjects received 1.8 mg liraglutide for 22 weeks. Administered subcutaneously (s.c., under the skin) once daily.
- Liraglutide Placebo: Subjects randomised to 3 different placebo arms as an add-on to their pre-trial insulin treatment. Administered subcutaneously (s.c., under the skin) once daily. All the 3 arms were pooled together for data analysis.
  1. Placebo 0.1 mL arm: Subjects received 0.1 mL placebo throughout the trial.
  2. Placebo 0.2 mL arm: Subjects received 0.1 mL placebo for 2 weeks followed by 0.2 mL for 24 weeks.
  3. Placebo 0.3 mL arm: Subjects received 0.1 mL placebo for 2 weeks followed by 0.2 mL for 2 weeks and 0.3 mL for next 22 weeks of the trial period.
Period: Overall Study
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Started | 212 | 209 | 207 | 207
Exposed | 211 | 209 | 206 | 206
Completed | 186 | 177 | 165 | 180
Not Completed | 26 | 32 | 42 | 27
Not completed — Protocol Violation | 2 | 2 | 0 | 7
Not completed — Withdrawal by Subject | 10 | 10 | 5 | 13
Not completed — Adverse Event | 12 | 19 | 34 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0 | 3
Not completed — Unclassified | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Baseline (BL) characteristics were presented for full analysis set (FAS = 831 subjects). Out of 835 randomised subjects, 4 were excluded from FAS:1 subject each in the lira 1.8 mg, 0.6 mg and placebo arm were not exposed to trial treatment and 1 subject in the lira 1.8 mg arm had no post-BL measurements.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Liraglutide Placebo | Total
Number analyzed (Participants) | 211 | 209 | 205 | 206 | 831
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (12.88) | 42.8 (13.31) | 43.2 (12.9) | 42.7 (12.97) | 43.2 (13.00)
Gender [Count of Participants; unit: Participants]
  Female | 118 | 106 | 113 | 112 | 449
  Male | 93 | 103 | 92 | 94 | 382
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 8.09 (0.743) | 8.07 (0.731) | 8.04 (0.736) | 8.12 (0.723) | 8.08 (0.732)
Body Weight [Mean (Standard Deviation); unit: kg] | 83.10 (16.137) | 84.69 (18.155) | 83.64 (17.620) | 84.20 (16.539) | 83.91 (17.109)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in glycosylated haemoglobin (HbA1c), after 26 weeks of treatment. Full analysis set (FAS = 831) included all randomised subjects who had received at least one dose and had any post-randomisation data.
Time Frame: Week 0, Week 26
Population: Out of the 831 subjects in FAS, 22 subjects in lira 0.6 mg arm, 33 subjects in lira 1.2 mg arm, 35 subjects in lira 1.8 mg arm and 16 in placebo arm did not contribute to this analysis. Missing data imputed from a mixed model for repeated measurements (MMRM) method.
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 189 | 176 | 170 | 190
Percent (%) glycosylated haemoglobin | -0.23 (0.744) | -0.23 (0.731) | -0.32 (0.73) | 0.01 (0.674)
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; Superiority of liraglutide 1.8 mg versus placebo was planned to be concluded if and only if the upper limit of the two-sided 95% confidence interval for the estimated difference in HbA1c was less than zero; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.5 to -0.2]
Statistical Analysis 2: Comparison: Liraglutide 1.2 mg vs Liraglutide Placebo; Superiority of liraglutide 1.2 mg was planned to be evaluated only if superiority for liraglutide 1.8 mg was concluded; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.38 to -0.08]
Statistical Analysis 3: Comparison: Liraglutide 0.6 mg vs Liraglutide Placebo; Superiority of liraglutide 0.6 mg versus placebo was planned to be evaluated only if superiority of liraglutide 1.2 mg was concluded; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.39 to -0.1]

2. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline body weight, after 26 weeks of treatment. Full analysis set (FAS = 831) included all randomised subjects who had received at least one dose and had any post-randomisation data.
Time Frame: Week 0, Week 26
Population: Of the 831 subjects in FAS, 27 subjects in lira 0.6 mg arm, 38 subjects in lira 1.2 mg arm, 35 subjects in lira 1.8 mg arm and 26 in placebo arm did not contribute to the analysis. Missing data imputed from a mixed model for repeated measurements (MMRM) method.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 184 | 171 | 170 | 180
kg | -2.37 (3.015) | -4.03 (3.677) | -5.1 (3.787) | -0.26 (2.782)

3. Secondary Outcome: Number of Treatment-emergent Symptomatic Hypoglycaemic Episodes
Description: Number of treatment-emergent symptomatic hypoglycaemic episodes during 26 weeks of treatment. Symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification or a self-measured plasma glucose (SMPG) value of <3.1 mmol/L (56 mg/dL), with symptoms consistent with hypoglycaemia. Severe hypoglycaemia as per ADA classification is defined as an episode that required assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions.
Time Frame: Weeks 0-26
Population: Safety analysis set (SAS) included all subjects exposed to at least one dose of randomised liraglutide or placebo (SAS = 832 subjects). Symptomatic hypoglycaemic episodes were reported by 166 subjects in liraglutide 0.6 mg arm, 175 subjects in liraglutide 1.2 mg, 160 subjects in liraglutide 1.8 mg arm and 162 subjects in liraglutide placebo arm.
Measure: Number; unit: episodes
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 211 | 209 | 206 | 206
episodes | 1437 | 1943 | 1490 | 1567

ADVERSE EVENTS:
Time Frame: From the first day of exposure to randomised treatment (week 0) to 7 days after the last day of randomised treatment (week 26).
Description: Safety analysis set (SAS) included all subjects exposed to at least one dose of randomised liraglutide or placebo.
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Serious Adverse Events (participants affected / at risk) | 20/211 | 21/209 | 14/206 | 14/206
Other Adverse Events (participants affected / at risk) | 137/211 | 164/209 | 162/206 | 125/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 0.6 mg (N=211) | Liraglutide 1.2 mg (N=209) | Liraglutide 1.8 mg (N=206) | Liraglutide Placebo (N=206)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (6) | 2 (2) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 3 (5) | 6 (7) | 2 (2) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 0.6 mg (N=211) | Liraglutide 1.2 mg (N=209) | Liraglutide 1.8 mg (N=206) | Liraglutide Placebo (N=206)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4) | 14 (18) | 7 (7) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8) | 8 (13) | 14 (17) | 5 (5)
Constipation (Gastrointestinal disorders) | 6 (6) | 23 (29) | 14 (15) | 9 (12)
Diarrhoea (Gastrointestinal disorders) | 14 (17) | 25 (30) | 30 (43) | 17 (22)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 19 (23) | 24 (35) | 1 (1)
Nausea (Gastrointestinal disorders) | 68 (81) | 97 (122) | 102 (170) | 34 (40)
Vomiting (Gastrointestinal disorders) | 19 (25) | 29 (40) | 35 (65) | 7 (8)
Fatigue (General disorders) | 13 (13) | 17 (18) | 22 (25) | 3 (5)
Gastroenteritis (Infections and infestations) | 6 (7) | 11 (11) | 8 (9) | 6 (6)
Influenza (Infections and infestations) | 15 (15) | 18 (23) | 18 (19) | 17 (20)
Nasopharyngitis (Infections and infestations) | 44 (59) | 40 (52) | 47 (67) | 46 (56)
Sinusitis (Infections and infestations) | 7 (7) | 11 (12) | 3 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 14 (20) | 11 (13) | 11 (14) | 25 (31)
Decreased appetite (Metabolism and nutrition disorders) | 21 (21) | 40 (42) | 50 (55) | 9 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (14) | 13 (17) | 12 (16) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (6) | 8 (10) | 14 (15)
Headache (Nervous system disorders) | 16 (27) | 26 (33) | 30 (43) | 30 (40)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 4 (4) | 14 (19) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to Novo Nordisk before submission for comments. Comments will be given within four weeks from receipt of the planned communication.